CLINICAL TRIAL: NCT00002878
Title: A PHASE III STUDY OF PSC-833 IN COMBINATION WITH VINCRISTINE, DOXORUBICIN AND DEXAMETHASONE (PSC-833/VAD) VERSUS VAD ALONE IN PATIENTS WITH RELAPSING OR REFRACTORY MULTIPLE MYELOMA
Brief Title: Combination Chemotherapy With or Without PSC 833 in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065178; E-1A95; CAN-NCIC-MY8; CLB-E1A95; EORTC-E1A95/06971; SWOG-E1A95; CAN-NCIC-J1A95; CLB-9596; SWOG-S1A95
Record Dates: First submitted 1999-11-01; First posted 2003-07-09 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Doxorubicin; valspodar; Vincristine

INTERVENTIONS:
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: valspodar
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Some tumors become resistant to chemotherapy drugs. Combining PSC 833 with chemotherapy may reduce resistance to the drug, and allow more tumor cells to be killed. It is not yet known whether combination chemotherapy plus PSC 833 is more effective than combination chemotherapy alone in treating patients with relapsed or refractory multiple myeloma.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without PSC 833 in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and objective response rate of patients with relapsed or refractory multiple myeloma treated with vincristine, doxorubicin, and dexamethasone (VAD) with or without PSC 833.
* Compare event free survival and subjective response in patients treated with these regimens.
* Correlate treatment outcome with p-glycoprotein expression.
* Determine whether prognostic factors previously determined to be useful in untreated patients (i.e., plasma cell labeling index and multidrug resistance determined from bone marrow aspirates, serum beta 2-microglobulin and interleukin-6 receptor levels) correlate with objective and subjective response and event-free and overall survival in patients treated with these regimens.
* Compare the toxicity of VAD with or without PSC 833.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by response to prior treatment, prior doxorubicin and/or vincristine, prior autologous peripheral blood stem cell transplantation, and center.

Patients are randomized to 1 of 2 treatment arms:

* Arm I: The first group receives vincristine, doxorubicin, and dexamethasone (VAD). Patients receive higher dose vincristine IV over 96 hours and higher dose doxorubicin IV over 96 hours on days 1-4 and oral dexamethasone daily on days 1-4 and 15-18.
* Arm II: The second group receives VAD plus oral PSC 833. Patients receive oral PSC 833 every 6 hours beginning on day 1 and continuing for 20 doses. Patients receive lower dose vincristine IV over 96 hours and lower dose doxorubicin IV over 96 hours on days 2-5 and oral dexamethasone daily on days 2-5 and 16-19.

Treatment in both arms repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. After completion of 2 courses, patients are reevaluated, and those with stable or responding disease continue treatment for 2 courses beyond maximum response. Doxorubicin is discontinued in patients who receive a maximum lifetime dose but still have stable or responding disease.

Patients are followed every 2 months for survival.

PROJECTED ACCRUAL: A total of 360 patients will be accrued for this study over approximately 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Multiple myeloma of any stage confirmed by:

  * Bone marrow plasmacytosis with at least 10% plasma cells, sheets of plasma cells, or biopsy proven plasmacytosis
  * Myeloma (M) protein in serum and/or urine
* Measurable disease by at least one of the following:

  * Serum M-component at least 1.0 g/dL by electrophoresis

    * Baseline measurement by nephelometry also, if used to follow response
  * Urine M-protein excretion greater than 200 mg/24 hours by electrophoresis
* The following are not considered measurable but are followed for response:

  * Lytic bone lesions
  * Bone marrow plasmacytosis
  * Anemia
  * Serum beta 2-microglobulin
* Objective evidence of progression by at least one of the following:

  * Increased serum M-protein (by electrophoresis unless M-spike less than 1.5 g/dL)

    * At least 50% above lowest remission level or by at least 2 g/dL
    * To more than 1.0 g/dL if sole protein indication of relapse
    * Nephelometry may be used instead of electrophoresis
  * Increased urine M-protein

    * To 50% above lowest level OR by 2 g/24 hours
    * To greater than 200 mg/24 hours
  * Definite new lytic bone lesions or at least a 50% increase in size of existing lesions (discussion with ECOG Study Chairman required if sole indication of progression)
  * Increase in serum or urine M-protein by 25% to under 50% (as above) plus one of the following:

    * Serum calcium greater than 12 mg/dL without other cause
    * Hemoglobin decreased by more than 2.0 g/dL not attributed to chemotherapy, interferon therapy, or a myelodysplastic syndrome

      * Less than 11 g/dL in men
      * Less than 10 g/dL in women
    * At least a 50% increase in bone marrow plasmacytosis
* Failure of prior cytotoxic therapy defined by one of the following:

  * Never responded
  * Relapsed within 2 months of last treatment
  * Relapsed 2-12 months after last treatment following initial response
* Adequate prior chemotherapy required, e.g.:

  * At least 2 courses of combination chemotherapy (e.g., VBMCP, VBAP, MP)

    * Prior vincristine, doxorubicin, and dexamethasone (VAD) allowed

      * No demonstrated resistance to VAD
      * At least 3 months since prior VAD
    * Cumulative doxorubicin dose no more than 250 mg/m2
    * Prior autologous peripheral blood stem cell transplant allowed if performed prior to development of drug resistance

      * No prior allogeneic transplant
* No smoldering myeloma, localized plasmacytoma, or monoclonal gammopathy of undetermined significance (MGUS)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-3

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST less than 1.5 times ULN
* No chronic or active hepatitis or cirrhosis

Renal:

* Creatinine less than 3.0 mg/dL

Cardiovascular:

* Ejection fraction at least 50%
* No history of congestive heart failure
* No overt angina despite medication
* No myocardial infarction within 2 months
* No poorly controlled hypertension (i.e., pressure 200/110 or higher despite medication)
* No arrhythmia requiring therapy (i.e., sustained atrial or ventricular arrhythmia or multifocal premature ventricular contraction)

  * Digoxin to control ventricular rate of atrial fibrillation that has been chronic for more than 1 month allowed

Neurologic:

* No peripheral neuropathy with weakness
* No cerebellar disease with ataxia

Gastrointestinal:

* Adequate gastrointestinal function to allow absorption of PSC 833
* No active peptic ulcer

Other:

* No hypersensitivity to PSC 833 or cyclosporine
* No active infection
* HIV negative
* No uncontrolled diabetes mellitus
* No second malignancy within the past 5 years except curatively treated nonmelanomatous skin cancer, carcinoma in situ of the cervix, or other localized cancer treated with surgery alone
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious medical problem unless sufficiently stabilized

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic therapy (e.g., interferon) allowed

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since other prior chemotherapy (including plicamycin)

Endocrine therapy:

* At least 2 weeks since high dose steroids (at least 100 mg/m2/day of prednisone or at least 40 mg/day of dexamethasone (including steroids for hypercalcemia)

Radiotherapy:

* At least 2 weeks since prior radiotherapy except limited radiotherapy to a single bone lesion

Surgery:

* At least 4 weeks since prior major surgery

Other:

* No concurrent anticoagulants
* No concurrent drugs known to modulate cyclosporine blood concentrations

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-06-30 (Actual); Primary Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R. Friedenberg, MD, Study Chair — Guthrie Cancer Center at Guthrie Clinic Sayre; Karl H. Hanson, MD, Study Chair — Saint Luke's Cancer Institute at Saint Luke's Hospital; Richard A. Larson, MD, Study Chair — University of Chicago; Chaim Shustik, MD, Study Chair — Royal Victoria Hospital - Montreal; Pieter Sonneveld, MD, PhD, Study Chair — University Medical Center Rotterdam at Erasmus Medical Center
Locations (40):
- United States (32):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
- Canada (8):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec

REFERENCES:
- [Result] Friedenberg WR, Rue M, Blood EA, Dalton WS, Shustik C, Larson RA, Sonneveld P, Greipp PR. Phase III study of PSC-833 (valspodar) in combination with vincristine, doxorubicin, and dexamethasone (valspodar/VAD) versus VAD alone in patients with recurring or refractory multiple myeloma (E1A95): a trial of the Eastern Cooperative Oncology Group. Cancer. 2006 Feb 15;106(4):830-8. doi: 10.1002/cncr.21666. PMID 16419071